CLINICAL TRIAL: NCT04796272
Title: Role of Individualized Versus Traditional Exercise in Combating Fatigue in Fatigued Multiple Sclerosis Patients
Brief Title: Role of Individualized Versus Traditional Exercise in Combating Fatigue
Acronym: REEN-SEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low inclusion rates
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20CH032; 2020-A00841-38 (Other: IDRCB)
Record Dates: First submitted 2021-01-15; First posted 2021-03-12 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; individual exercise; fatigue; traditional exercise
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Acclimatization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional exercise (Active Comparator): fatigued multiple sclerosis patients with a traditional training program
  Interventions: Other: traditional training program
- Individual exercise (Experimental): tired multiple sclerosis patients with an adapted and individualized training program
  Interventions: Other: Adapted and individualized physical training program

INTERVENTIONS:
Other: Adapted and individualized physical training program — Physical training program adapted and individualized according to each patient in this group
  Arms: Individual exercise
Other: traditional training program — Same training program for all patients in this group
  Arms: Traditional exercise

SUMMARY:
The objective of this project will be to characterise the benefits of an exercise programme adapted to each individual's abilities compared to a traditional exercise programme with the aim of reducing perceived fatigue and improving the quality of life of Patients with multiple sclerosis.

DETAILED DESCRIPTION:
Chronic fatigue is a very common symptom reported (80%) by patients with multiple sclerosis (MS), regardless of the type of MS and level of disability. Despite the clinical importance of MS-related fatigue, pharmacological treatments remain quite ineffective in preventing or treating chronic fatigue.

Recently, physical activity has proven to be an effective therapy with benefits on chronic fatigue as well as on different functions (muscular, cardiorespiratory, cognitive, etc.). Nevertheless, the effects of physical exercise may vary between MS patients, as MS is a heterogeneous disease and does not affect each individual in the same way. The objective of this project will be to characterise the benefits of an exercise programme adapted to each individual's abilities compared to a traditional exercise programme with the aim of reducing perceived fatigue and improving the quality of life of Patients with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70 years old
* Male or female
* With relapsing-remitting multiple sclerosis (RRMS) as defined by McDonald's 2010 criteria.
* Between 2 and 25 years from the onset of multiple sclerosis
* With a high level of fatigue, corresponding to a score of Fatigue Severity Scale> 4 and Fatigue questionnaire > 38.
* Expanded Disability Status Scale Score 5
* Testing ≥ 4 in all leg muscles.
* Ability to walk for 10 minutes without stopping (self-reported)
* Affiliates or beneficiaries of a social security scheme
* Having freely given their written consent after having been informed of the purpose, course of action and potential risks involved

Exclusion Criteria:

* Severe cerebellar spasticity or ataxia in either leg.
* Abnormal range of motion of the toes and/or ankle.
* Musculoskeletal injury that interferes with pedaling.
* High resting heart rate (>90 beats per minute).
* Blood pressure > 144/94 mmHg.
* Onset of a multiple sclerosis attack within 90 days prior to the study.
* Recent adjustment of any medication or drugs that may impact on fatigue, or taking stimulants for fatigue (e.g. Modafinil).
* Taking of neuro-active substances that may impair cortico-spinal excitability (hypnotics, antiepileptics, psychotropic drugs, muscle relaxants) throughout the study period.
* Contraindication to the application of a magnetic field
* History of co-morbid disease or conditions that would compromise the subject's safety during the study.
* Participation at the same time in another medical intervention study or having participated in such a study within 30 days prior to this study.
* Pregnant and Nursing Women
* Women of childbearing age without effective contraception
* Patient unable to understand the purpose and conditions of the study, incapable of giving consent
* Patient deprived of liberty or patient under guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Chronic fatigue score | Month 3
  assessed using the Fatigue Severity Scale (FSS) questionnaire before and after an individualized re-training program compared to a traditional re-training program in MS patients.

SECONDARY OUTCOMES:
cardiorespiratory fitness | Month 3
  evaluated by measuring the maximum oxygen consumption (VO2max) during an incremental exercise on a cycloergometer.
Hematological parameters | Month 3
  red blood cell and hemoglobin levels measured by spectrophotometry.
Inflammatory parameters | Month 3
  c-reactive protein
quality of sleep | Month 3
  actigraphy measurements and sleep diary records
cortical activation level | Month 3
  transcranial magnetic stimulation
cortico-spinal excitability | Month 3
  transcranial magnetic stimulation
neuromuscular fatigue of peripheral function | Month 3
  electrical nerve stimulation
Analysis overall quality of life : Fatigue questionnaire | Month 3
  Fatigue questionnaire by Modified Fatigue Impact Scale (MFIS) results
Analysis overall quality of life :Quality of Life | Month 3
  Quality of Life Questionnaire by SEP-59 results
Analysis overall quality of life :Depression | Month 3
  Depression Questionnaire by Center for Epidemiologic Studies Depression (CES-D) results
Analysis overall quality of life : Sleep Quality | Month 3
  Sleep Quality Questionnaire by Pittsburgh Sleep Quality Index (PSQ-I) results
Analysis overall quality of life : Physical Activity | Month 3
  Physical Activity Questionnaire by Godin Leisure-Time Exercise Questionnaire (GLTEQ) results

CONTACTS AND LOCATIONS:
Overall Officials: Jean Philippe CAMDESSANCHE, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No